CLINICAL TRIAL: NCT00221156
Title: Effects of Acarbose Long-Term Therapy on Prevention of Cardiovascular Events in Abnormal Glucose Tolerance With Coronary Artery Disease (ALERT Study)
Brief Title: Acarbose and Secondary Prevention After Coronary Stenting
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Translational Research Center for Medical Innovation, Kobe, Hyogo, Japan (Other)
Collaborators: Institute of Biomedical Research and Innovation, Kobe, Hyogo, Japan (Other); Kobe City General Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: BRI_CAD_04-02
Record Dates: First submitted 2005-09-13; First posted 2005-09-22 (Estimated); Last update posted 2009-06-25 (Estimated); Status verified 2009-06

CONDITIONS: Glucose Metabolism Disorders; Coronary Artery Disease
Keywords: Abnormal Glucose Tolerance; coronary artery disease; diabetes mellitus; clinical outcome
MeSH Terms: conditions — Glucose Metabolism Disorders; Coronary Artery Disease; Diabetes Mellitus | interventions — Acarbose

INTERVENTIONS:
Drug: Acarbose

SUMMARY:
The purpose of this study is to determine whether the intervention for newly diagnosed abnormal glucose tolerance after coronary stenting will improve the long-term clinical outcome.

DETAILED DESCRIPTION:
Recent studies have demonstrated that newly diagnosed abnormal glucose tolerance (AGT; diabetes mellitus and impaired glucose tolerance) are common among the patients with ischemic heart disease. Several large cohort studies indicate that people with prediabetic conditions, such as impaired glucose tolerance, have a raised risk of future cardiovascular disease. Intervention with acarbose can prevent myocardial infarction and cardiovascular disease in type 2 diabetic and IGT patients. However, the effect of acarbose to secondary prevention of myocardial infarction or cardiovascular events in patients with newly diagnosed AGT after coronary stenting remains unclear. The purpose of the present study is to determine whether the intervention to such abnormalities after coronary stenting will improve the long-term clinical outcome. This is a opened, randomized study to compare acarbose versus a standard lifestyle modification. Patients will have a 1:1 chance of receiving acarbose versus the standard lifestyle modification. There is some research evidence that suggests acarbose may improve clinical outcome in patients with type 2 diabetes and in IGT patients.

ELIGIBILITY:
Inclusion Criteria:

* Within 8 weeks since implantation of coronary artery stents for stable angina pectoris or acute coronary syndrome.
* Abnormal glucose tolerance according to a 75 g oral glucose tolerance test (OGTT).
* HbA1c is less than 6.5%.
* Age is between 20 and 75 years (at time of consent).
* Patients who can give informed consent themselves in writing.

Exclusion Criteria:

* Patients with abnormal glucose tolerance caused by other organic disorders such as pancreatitis, hemochromatosis, post pancreatectomy, hyperthyroidism, Cushing syndrome, Prader-Willi syndrome, etc.
* Patients with planned angioplasty.
* Patients with uncontrollable congestive heart failure.
* Less than 6 months since last episode of cerebral infarction.
* Patients who have received medication for diabetes mellitus before.
* AST (GOT) exceeding 100 IU/L or ALT (GPT) exceeding 100 IU/L.
* Creatinine exceeding 2 mg/dl.
* Patients with a history of ileus or less than 6 months since celiotomy.
* Pregnant women or those who plan to become pregnant, or are in the lactation period.
* Habitual drinker (more than 100 ml/day of alcohol).
* Patients with a history of gastrectomy.
* Patients for whom it is impossible to follow up for 5 years.
* Any other reason that the clinical supervisors or clinical researchers may have for considering a case unsuitable for the study.

Ages: 20 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2005-05; Study Completion 2009-04 (Actual)

PRIMARY OUTCOMES:
Cardiovascular event free survival time

SECONDARY OUTCOMES:
Conversion of abnormal glucose tolerance to type 2 diabetes
All causes of death
Occurrence of every cardiovascular event
Occurrence of in-stent restenosis
Change in fasting, 2-hour blood glucose and insulin level
Change in homeostasis model assessment of insulin resistance
Change in hemoglobin A1c (HbA1c)
Change in lipid profile

CONTACTS AND LOCATIONS:
Overall Officials: Koichi Tamita, MD., Principal Investigator — Division of Cardiology, Kobe General Hospital; Minako Katayama, MD, Study Director — Division of Clinical Research Promotion, Institute of Biomedical Research and Innovation.; Yutaka Furukawa, MD, Study Director — Division of Cardiology, Kobe General Hospital
Locations (3):
- Japan (3):
  - Institute of Biomedical Research and Innovation., Kobe, Hyogo Pref.
  - Kobe City General Hospital/Institute of Biomedical Research and Innovation, Kobe, Hyogo Pref.
  - Kawasaki Medical School Hospital, Kurashiki, Okayama-ken